CLINICAL TRIAL: NCT03238235
Title: A Randomised, Double Blind, Placebo Controlled Study to Evaluate the Micro-macroscopic Effects on Muscles, the Safety and Tolerability, and the Efficacy of Givinostat in Patients With Becker Muscular Dystrophy (BMD)
Brief Title: Clinical Study to Evaluate the Efficacy and Safety of Givinostat in Ambulant Patients With Becker Muscular Dystrophy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Italfarmaco (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DSC/15/2357/53; 2017-001629-41 (EudraCT Number)
Record Dates: First submitted 2017-07-12; First posted 2017-08-03 (Actual); Results first posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-03

CONDITIONS: Becker Muscular Dystrophy
Keywords: Givinostat; Becker Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — givinostat; givinostat hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo was indistinguishable from the active product in color, appearance, smell and taste. Personnel involved in the study (Investigators, nurses, all other site personnel, clinical research associates [CRA], medical monitors, project managers, data managers and statisticians) were blinded at all times unless knowledge of the study treatment was necessary for the patient's safety.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Givinostat (Experimental): Givinostat oral suspension (10 mg/mL) twice daily in a fed state
  Interventions: Drug: Givinostat
- Placebo (Placebo Comparator): Placebo oral suspension (10 mg/mL) twice daily in a fed state
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Givinostat — suspension of Givinostat (10 mg/mL)
  Other Names: ITF2357
  Arms: Givinostat
Drug: Placebo — suspension manufactured to mimic Givinostat
  Other Names: Placebo Comparator: placebo
  Arms: Placebo

SUMMARY:
Objectives:

Primary objective: to establish the histological effects of Givinostat versus placebo administered over 12 months.

Secondary Objectives:

* To establish the macroscopic muscle effects of Givinostat versus placebo administered over 12 months assessed by Magnetic Resonance Imaging (MRI)/Magnetic Resonance Spectroscopy (MRS).
* To determine the other histological effects of Givinostat versus placebo administered over 12 months.
* To establish the efficacy of Givinostat versus placebo administered chronically over 12 months in slowing disease progression.
* To assess the safety and tolerability of Givinostat versus placebo administered chronically.
* To evaluate the pharmacokinetic (PK) profile of Givinostat administered chronically in the target population.
* To evaluate the impact of Givinostat versus placebo administered chronically on quality of life and activities of daily living.

DETAILED DESCRIPTION:
This was a phase 2, randomised, double-blind, placebo-controlled study. Eligible patients were randomized in a 2:1 ratio to receive Givinostat or placebo for 12 months. Randomization was stratified by concomitant steroid use at baseline (yes or no). The study comprised twelve (12) visits: screening (V1, V2), randomization (V3), treatment (V4-V10), end of study (V11) and follow-up (V12). Visits during treatment took place every 12 weeks, except for the first 2 months, when they occurred every 2 weeks to allow closer monitoring of safety.

Givinostat (ITF2357) oral suspension (10 mg/mL) was initially administered as 2 daily doses of 40-70 mg according to body weight after a meal (high dose). With amendment 2 of the protocol, a lower starting dose was implemented to address cases of thrombocytopenia reported following the treatment of the first 21 patients and corresponded to the reduced dose of the original protocol (i.e., 26.7-46.7 mg b.i.d according to body weight, i.e., low dose).

51 patients were to be enrolled to provide a sample size of 48 patients with evaluable baseline biopsies. Seventy patients provided written informed consent, 51 (72.86%) completed screening successfully and were randomized; 34 patients (66.67%) to the Givinostat group and 17 (33.33%) to the placebo group.

ELIGIBILITY:
Inclusion Criteria:

1. Ambulant patients with BMD diagnosis confirmed by genetic testing.
2. Able and willing to give informed consent in writing.
3. Able to perform 6MWT at screening with a minimum distance of 200 m and maximum distance of 450 m.
4. If in treatment with systemic corticosteroids and/or angiotensin-converting-enzyme (ACE) inhibitor , and/or β or α adrenergic receptor blocker, no significant change in dosage or dosing regimen (excluding changes related to body weight) was to be presented for a minimum of 6 months prior to start of study treatment.
5. Patients had to be willing to use adequate contraception from randomization until 3 months after the last dose of study treatment, and included the following:

   * True abstinence when in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar ovulation, symptothermal, post ovulation methods) and withdrawal were not acceptable methods of contraception.
   * Condom with spermicide, with the female partner using an acceptable method of contraception, such as an oral, transdermal, injectable or implanted steroid-based contraceptive, or a diaphragm or a barrier method of contraception in conjunction with spermicidal jelly such as a cervical cap with spermicide jelly.

Exclusion Criteria:

1. Exposure to another investigational drug within 3 months prior to the start of study treatment.
2. Use of any pharmacological treatment, other than corticosteroids, that could have affected muscle strength or function within 3 months prior to the start of study treatment (e.g., growth hormone). vitamin D, calcium, and other supplements were allowed.
3. Surgery that could have affected muscle strength or function within 3 months before study entry or planned surgery at any time during the study.
4. Presence of other clinically significant disease that in the Investigator's opinion could have adversely affected the safety of the patient or could have impaired the assessment of study results.
5. A diagnosis of other uncontrolled neurological diseases or presence of relevant somatic disorders not related to BMD that could have interfered with the ability to perform the muscle function tests and/or to comply with the study protocol procedures.
6. Platelet count, white blood cell (WBC) count and hemoglobin at screening less than the lower limit of normal (LLN). If laboratory screening results were < LLN, platelet count, WBC count and hemoglobin were to be repeated once, and if again < LLN became exclusionary.
7. Symptomatic cardiomyopathy or heart failure (New York Heart Association Class III or IV) or left ventricular ejection fraction < 50% at screening or with heart transplant.
8. Current liver disease or impairment, including but not limited to elevated total bilirubin (>. 1.5 x upper limit of normal [ULN]), unless secondary to Gilbert's disease or pattern consistent with Gilbert's disease.
9. Inadequate renal function defined by serum cystatin C > 2 x ULN. If the value was > 2 x ULN, serum Cystatin C was to be repeated once, and if again > 2 x ULN became exclusionary.
10. Positive test for hepatitis B surface antigen, hepatitis C antibody, or human immunodeficiency virus at screening.
11. Baseline corrected QT interval using Fridericia's correction (QTcF) > 450 msec (as the mean of 3 consecutive readings 5 minutes apart) or history of additional risk factors for torsades de pointes (e.g., heart failure, hypokalemia, or family history of long QT syndrome).
12. Current psychiatric illness/social situations rendering the patient unable to understand or comply with the muscle function tests and/or with the study protocol procedures.
13. Hypersensitivity to the components of the study medication.
14. Sorbitol intolerance or sorbitol malabsorption, or the hereditary form of fructose intolerance.
15. Contraindications for muscle biopsy.
16. Contraindications forMRI/MRS (e.g., claustrophobia, metal implants or seizure disorders).
17. Hypertriglyceridemia (˃ 1.5 x ULN). At screening, patients with hypertriglyceridemia could be enrolled if on stable treatment and with controlled levels of triglycerides (i.e., within normal range) for at least six months.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2018-01-09 (Actual); Primary Completion 2021-03-19 (Actual); Study Completion 2021-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giacomo Comi, MD, Principal Investigator — Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico di Milano
Locations (2):
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico di Milano, UOS, Milan, Italy
- Leiden University Medical Center LUMC, Leiden, Netherlands

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Seventy patients provided written informed consent to participate in this study. Fifty-one patients (72.86%) completed screening successfully and were randomized; 34 patients (66.67%) were assigned to the Givinostat group and 17 (33.33%) to the placebo group.
Period: Overall Study
Arm/Group | Givinostat | Placebo
Started | 34 | 17
Per Protocol | 25 | 14
ITT | 34 | 17
Safety | 34 | 17
PK | 34 | 17
Completed | 30 | 17
Not Completed | 4 | 0
Not completed — Adverse Event | 2 | 0
Not completed — patients unable to travel to the site due to the COVID-19 pandemic | 2 | 0

BASELINE CHARACTERISTICS:
Population: Intent-To-Treat Analysis (ITT) Set: all patients assigned treatment by randomization who received at least one dose of study medication. According to the intent to treat principle, patients were analyzed according to the treatment assigned. Efficacy analyses were performed on the ITT set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Givinostat | Placebo | Total
Number analyzed (Participants) | 34 | 17 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 17 | 51
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.5 (11.56) | 39.2 (9.84) | 37.4 (10.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 34 | 17 | 51
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 17 | 18
  White | 33 | 0 | 33
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Netherlands | 3 | 3 | 6
  Italy | 31 | 14 | 45

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline to Visit 11 in Total Fibrosis (%) on Log Scale, Comparing the Histology of Muscle Biopsies
Description: The primary efficacy assessment was the mean total fibrosis (%) on log scale assessed through histological examination of bicep muscle biopsies at two timepoints (At baseline and at Visit 11). More particularly, patients underwent two biopsies of muscle from the brachial biceps: the first before starting the study treatment (Visit 2, baseline), and the second at the end of treatment (Visit 11). For each patient, the percentage of total fibrosis was calculated as log of the least square mean of the available fields at each evaluation.
Time Frame: after 12 months of treatment (at Visit 11)
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: log[percentage of total fibrosis]
Units Other Than Participants: # fields for each biopsy sample
Arm/Group | Givinostat | Placebo
Number analyzed (Participants) | 29 | 15
Number analyzed (# fields for each biopsy sample) | 4 | 4
log[percentage of total fibrosis] | -0.017 [-0.367 to 0.333] | -0.054 [-0.507 to 0.399]
Statistical Analysis 1: Comparison: Givinostat vs Placebo; total fibrosis at visit 11; Test type: Superiority; p = 0.8282, ANCOVA — ANCOVA model was performed considering the difference between log of total fibrosis and log baseline values as dependent variable; log baseline value was included as covariate, treatment and concomitant steroid use as independent class variables; Log Difference of the least square means = 0.04, 95% CI 2-sided [-0.30 to 0.38]
Statistical Analysis 2: Comparison: Givinostat vs Placebo; A Mixed Model was fitted to the data in order to evaluate the difference in total fibrosis between biopsy sites; Test type: Superiority — Mixed model was performed considering the difference between log Visit 11 and log baseline values as dependent variable; log baseline as covariate, treatment was included as independent class variable and treatment by sequence interaction. The sequence of biopsy site (R-L, L-R) was included as a fixed effect and subject as a random effect. If the treatment by sequence interaction was p>0.10, then the model without the interaction term is presented; p = 0.6465, Mixed Models Analysis; Log Difference of Least Square Means = -0.11, 95% CI 2-sided [-0.59 to 0.37]

2. Secondary Outcome: Mean Change From Baseline to Visit 11 in the Percentage of Fat Fraction of Vastus Lateralis and Soleus
Description: Evaluation was performed comparing Magnetic Resonance Spectroscopy (MRS) before and after 12 months of treatment with Givinostat versus placebo. Please note that Statistics data are expressed as log least square mean (IC 95%) for the vastus lateralis and as least square mean (IC 95%) back-transformed on the original scale for the soleus.
Time Frame: after 12 months of treatment (at Visit 11)
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: log[percentage of fat in muscle]
Units Other Than Participants: muscle images for timepoint
Arm/Group | Givinostat | Placebo
Number analyzed (Participants) | 34 | 17
Number analyzed (muscle images for timepoint) | 1 | 1
log[percentage of fat in muscle]
  Vastus Lateralis: number analyzed (Participants) | 33 | 17
  Vastus Lateralis | 0.017 [-0.053 to 0.086] | 0.064 [-0.019 to 0.147]
  Soleus: number analyzed (Participants) | 27 | 14
  Soleus | -4.287 [-6.126 to -2.447] | -4.021 [-6.404 to -1.637]
Statistical Analysis 1: Comparison: Givinostat vs Placebo; Vastus lateralis; Test type: Superiority; p = 0.1991, ANCOVA — ANCOVA model was performed considering baseline fat fraction of vastus lateralis or fat fraction in the soleus value as covariate and treatment and concomitant steroid use at baseline as independent class variables; Log Difference of Least Square Means = -0.05, 95% CI 2-sided [-0.12 to 0.03]
Statistical Analysis 2: Comparison: Givinostat vs Placebo; Soleus; Test type: Superiority; p = 0.7849, ANCOVA — [p-value comment as in outcome 2, analysis 1]; difference of the least square means = -0.27, 95% CI 2-sided [-2.22 to 1.69]

3. Secondary Outcome: Mean Change From Baseline to Visit 11 in the Percentage of Fat Fraction of Lower Limb Muscles
Description: Evaluation was performed comparing Dixon Magnetic Resonance Imaging (MRI) before and after 12 months of treatment with Givinostat versus placebo.
  The lower limb muscles assessed were: whole thigh, quadriceps, medial thigh, hamstrings, triceps surae and pelvic girdle. Please note that statistics data are expressed as: Least Square Means (95% CI) for whole thigh, quadriceps, hamstrings, triceps surae and pelvis girdle; while as Log Least Square Means (95% CI) for medial thigh.
Time Frame: after 12 months of treatment (at Visit 11)
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of fat in muscle
Units Other Than Participants: MRI images for each timepoint
Arm/Group | Givinostat | Placebo
Number analyzed (Participants) | 34 | 17
Number analyzed (MRI images for each timepoint) | 5 | 5
percentage of fat in muscle
  Whole Thigh: number analyzed (Participants) | 33 | 17
  Whole Thigh: number analyzed (MRI images for each timepoint) | 5 | 2
  Whole Thigh | 0.642 [-0.328 to 1.611] | 1.996 [0.813 to 3.180]
  Quadriceps: number analyzed (Participants) | 33 | 17
  Quadriceps: number analyzed (MRI images for each timepoint) | 5 | 2
  Quadriceps | 0.610 [-0.506 to 1.726] | 2.572 [1.227 to 3.918]
  Hamstrings: number analyzed (Participants) | 33 | 17
  Hamstrings: number analyzed (MRI images for each timepoint) | 5 | 2
  Hamstrings | 0.877 [-0.627 to 2.381] | 1.455 [-0.400 to 3.309]
  Triceps Surae: number analyzed (Participants) | 22 | 11
  Triceps Surae: number analyzed (MRI images for each timepoint) | 5 | 2
  Triceps Surae | -0.276 [-2.862 to 2.310] | 1.317 [-1.686 to 4.319]
  Pelvis Girdle: number analyzed (Participants) | 33 | 17
  Pelvis Girdle: number analyzed (MRI images for each timepoint) | 5 | 2
  Pelvis Girdle | 0.584 [-0.509 to 1.676] | 1.471 [0.112 to 2.830]
Statistical Analysis 1: Comparison: Givinostat vs Placebo; Whole thigh at visit 11; Test type: Superiority; p = 0.0149, ANCOVA — ANCOVA model was performed considering baseline Fat Fraction of lower limb muscles value as covariate and treatment and concomitant steroid use at baseline as independent class variables; Difference of Least Square Means = -1.35, 95% CI 2-sided [-2.43 to -0.28]
Statistical Analysis 2: Comparison: Givinostat vs Placebo; Quadriceps at visit 11; Test type: Superiority; p = 0.0022, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Difference of Least Square Means = -1.96, 95% CI 2-sided [-3.18 to -0.75]
Statistical Analysis 3: Comparison: Givinostat vs Placebo; Hamstrings at visit 11; Test type: Superiority; p = 0.4869, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Difference of least square means = -0.58, 95% CI 2-sided [-2.24 to 1.08]
Statistical Analysis 4: Comparison: Givinostat vs Placebo; Triceps Surae at Visit 11; Test type: Superiority; p = 0.0939, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Difference of Least Square Means = -1.59, 95% CI 2-sided [-3.47 to 0.29]
Statistical Analysis 5: Comparison: Givinostat vs Placebo; Pelvis girdle at visit 11; Test type: Superiority; p = 0.1579, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Difference of Least Square Means = -0.89, 95% CI 2-sided [-2.13 to 0.36]

4. Secondary Outcome: Mean Change From Baseline to Visit 11 in Cross-sectional Area (CSA), in cm2 of Lower Limb Muscles
Description: Evaluation was performed comparing Dixon MRI findings before and after 12 months of treatment with Givinostat versus placebo.
  Dixon technique has advantages in multiple applications for evaluation of musculoskeletal system diseases. It allows more robust fat suppression than do other sequences and can be used in combination with multiple different sequences (GRE and SE) and using different weightings (T1, T2, or proton density).
  The lower limb muscles assessed were: whole thigh, quadriceps, medial thigh, hamstrings, triceps surae and pelvic girdle (data showed as least square mean)
Time Frame: after 12 months of treatment (Visit 11)
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: centimeters^2
Units Other Than Participants: MRI images for each timepoint
Arm/Group | Givinostat | Placebo
Number analyzed (Participants) | 34 | 17
Number analyzed (MRI images for each timepoint) | 5 | 5
centimeters^2
  whole thigh: number analyzed (Participants) | 33 | 17
  whole thigh | 2.782 [0.151 to 5.413] | 2.377 [-0.820 to 5.575]
  quadriceps: number analyzed (Participants) | 33 | 17
  quadriceps | 0.997 [-0.169 to 2.163] | 1.082 [-0.329 to 2.494]
  medial thigh: number analyzed (Participants) | 33 | 17
  medial thigh | 0.669 [-0.468 to 1.807] | 0.321 [-1.060 to 1.702]
  hamstrings: number analyzed (Participants) | 33 | 17
  hamstrings | 1.103 [0.108 to 2.098] | 0.994 [-0.207 to 2.195]
  triceps surae: number analyzed (Participants) | 22 | 11
  triceps surae | -0.033 [-3.699 to 3.634] | 0.183 [-3.756 to 4.122]
  pelvic girdle: number analyzed (Participants) | 33 | 17
  pelvic girdle | 1.284 [-0.494 to 3.062] | 0.965 [-1.187 to 3.116]
Statistical Analysis 1: Comparison: Givinostat vs Placebo; Whole Thigh at visit 11; Test type: Superiority; p = 0.7770, ANCOVA — ANCOVA model was performed considering baseline CSA as covariate, treatment and concomitant steroid use at baseline as independent class variables; Difference of Least Square Means = 0.40, 95% CI 2-sided [-2.45 to 3.26]
Statistical Analysis 2: Comparison: Givinostat vs Placebo; Quadriceps at Visit 11; Test type: Superiority; p = 0.8926, ANCOVA — [p-value comment as in outcome 4, analysis 1]; Difference of Least Square Means = -0.09, 95% CI 2-sided [-1.35 to 1.18]
Statistical Analysis 3: Comparison: Givinostat vs Placebo; Medial Thigh at Visit 11; Test type: Superiority; p = 0.5720, ANCOVA — [p-value comment as in outcome 4, analysis 1]; Difference of Least Square Means = 0.35, 95% CI 2-sided [-0.88 to 1.58]
Statistical Analysis 4: Comparison: Givinostat vs Placebo; Hamstrings at Visit 11; Test type: Superiority; p = 0.8386, ANCOVA — [p-value comment as in outcome 4, analysis 1]; Difference of Least Square Means = 0.11, 95% CI 2-sided [-0.97 to 1.18]
Statistical Analysis 5: Comparison: Givinostat vs Placebo; Triceps Surae at Visit 11; Test type: Superiority; p = 0.8591, ANCOVA — [p-value comment as in outcome 4, analysis 1]; Difference of Least Square Means = -0.22, 95% CI 2-sided [-2.68 to 2.25]
Statistical Analysis 6: Comparison: Givinostat vs Placebo; Pelvis Girdle at Visit 11; Test type: Superiority; p = 0.7392, ANCOVA; Difference of Least Square Means = 0.32, 95% CI 2-sided [-1.60 to 2.24]

5. Secondary Outcome: Mean Change From Baseline to Visit 11 in Contractile Area of Lower Limb Muscles (MRI)
Description: A summary of mean change in the contractile area of lower limb muscles comparing MRI findings before and after 12 months of treatment in the ITT set is reported. The lower limb muscles considered are the same as the outcome 3. Please note that statistic data are expressed as Least Square Means (95% CI) except for Hamstrings which is expressed as Log Least Square Means.
Time Frame: after 12 months of treatment
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: centimeters^2
Units Other Than Participants: MRI muscle images for each timepoint
Arm/Group | Givinostat | Placebo
Number analyzed (Participants) | 34 | 17
Number analyzed (MRI muscle images for each timepoint) | 5 | 5
centimeters^2
  Contractile Area in the Whole Thigh: number analyzed (Participants) | 33 | 17
  Contractile Area in the Whole Thigh | 0.309 [-0.853 to 1.470] | -1.057 [-2.466 to 0.352]
  Contractile Area in the Quadriceps: number analyzed (Participants) | 33 | 17
  Contractile Area in the Quadriceps | 0.139 [-0.458 to 0.735] | -0.493 [-1.195 to 0.210]
  Contractile Area in the Medial Thigh: number analyzed (Participants) | 33 | 17
  Contractile Area in the Medial Thigh | 0.162 [-0.342 to 0.665] | -0.197 [-0.813 to 0.420]
  Contractile Area in the Triceps Surae: number analyzed (Participants) | 22 | 11
  Contractile Area in the Triceps Surae | -0.542 [-3.598 to 2.514] | -1.291 [-4.632 to 2.050]
  Contractile Area in the Pelvis Girdle: number analyzed (Participants) | 33 | 17
  Contractile Area in the Pelvis Girdle | 0.257 [-0.420 to 0.933] | -0.287 [-1.133 to 0.559]
Statistical Analysis 1: Comparison: Givinostat vs Placebo; Whole Thigh at Visit 11; Test type: Superiority; p = 0.0375, ANCOVA — ANCOVA model was performed considering baseline Contractile Area value as covariate, treatment and concomitant steroid use at baseline as independent class variables; Difference of Least Square Means = 1.37, 95% CI 2-sided [0.08 to 2.65]
Statistical Analysis 2: Comparison: Givinostat vs Placebo; Quadriceps at Visit 11; Test type: Superiority; p = 0.0528, ANCOVA — [p-value comment as in outcome 5, analysis 1]; difference of least square means = 0.63, 95% CI 2-sided [-0.01 to 1.27]
Statistical Analysis 3: Comparison: Givinostat vs Placebo; Medial Thigh at Visit 11; Test type: Superiority; p = 0.2012, ANCOVA — [p-value comment as in outcome 5, analysis 1]; Difference of Least Square Means = 0.36, 95% CI 2-sided [-0.20 to 0.91]
Statistical Analysis 4: Comparison: Givinostat vs Placebo; Triceps Surae at Visit 11; Test type: Superiority; p = 0.4676, ANCOVA — [p-value comment as in outcome 5, analysis 1]; Difference of Least Square Means = 0.75, 95% CI 2-sided [-1.33 to 2.83]
Statistical Analysis 5: Comparison: Givinostat vs Placebo; Pelvis Girdle at Visit 11; Test type: Superiority; p = 0.1549, ANCOVA — [p-value comment as in outcome 5, analysis 1]; Difference of Least Square Means = 0.54, 95% CI 2-sided [-0.21 to 1.30]

6. Secondary Outcome: Mean Change From Baseline to Visit 11 in Biopsy Histology Parameters: CSA by Type (I or II Fibers), Total CSA
Description: A summary of the mean change in cross-sectional area (CSA) by type after 12 months of treatment in the ITT set is reported. Please note that descriptive statistic data are expressed as Log Least Square Means (95% CI) for CSA type I fibers, and as Least Square Means (95% CI) for CSA type II fibers and Total CSA.
Time Frame: After 12 months of treatment (Visit 11)
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: micrometers^2
Units Other Than Participants: # fields for each biopsy sample
Arm/Group | Givinostat | Placebo
Number analyzed (Participants) | 34 | 17
Number analyzed (# fields for each biopsy sample) | 4 | 4
micrometers^2
  CSA type II fibers: number analyzed (Participants) | 33 | 17
  CSA type II fibers: number analyzed (# fields for each biopsy sample) | 2 | 2
  CSA type II fibers | -25.320 [-1438.395 to 1387.755] | 593.875 [-1177.854 to 2365.604]
  Total CSA: number analyzed (Participants) | 33 | 17
  Total CSA | 642.505 [-603.081 to 1888.092] | 1215.047 [-359.764 to 2789.857]
Statistical Analysis 1: Comparison: Givinostat vs Placebo; CSA Type II at Visit 11; Test type: Superiority; p = 0.3240, ANCOVA — ANCOVA model was performed considering baseline biopsy histological parameters (Slide III) value as covariate, treatment and concomitant steroid use at baseline as independent class variables; Difference of Least Square Means = -619.20, 95% CI 2-sided [-1872.37 to 633.98]
Statistical Analysis 2: Comparison: Givinostat vs Placebo; Total CSA at Visit 11; Test type: Superiority; p = 0.3070, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Difference of Least Square Means = -572.54, 95% CI 2-sided [-1690.73 to 545.64]

7. Secondary Outcome: Mean Change From Baseline to Visit 11 in Percentage for the Following Histology Parameters: Fibers With Nuclear Centralizations (%), Total Number of Fibers (%), Regenerative Fibers (%).
Description: Evaluation of histologic parameters such as Fiber with nuclear centralizations (%), Total number of fibers (%), and Regenerative fibers (%) were performed comparing muscle biopsies after 12 months of treatment with Givinostat. Please note that descriptive statistic data are expressed as log least square mean for Regenerative fibers (%), and total number of fibers (Slides I), while are expressed as least square mean for Fibers with nuclear centralizations (%) and total number of fibers (Slides II and III).
Time Frame: after 12 months of treatment (Visit 11)
Population: Intent-To-Treat Analysis (ITT) Set: all patients assigned treatment by randomization who received at least one dose of study medication. According to the intent to treat principle, patients were analyzed according to the treatment assigned.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of fibers
Units Other Than Participants: # fields for each biopsy sample
Groups:
- Placebo: Placebo oral suspension (10 mg/mL) twice daily in a fed state
  Placebo: suspension manufactured to mimic Pivinostat
Arm/Group | Givinostat | Placebo
Number analyzed (Participants) | 34 | 17
Number analyzed (# fields for each biopsy sample) | 4 | 4
percentage of fibers
  Fibers with nuclear centralizations: number analyzed (Participants) | 29 | 15
  Fibers with nuclear centralizations | 0.196 [-0.183 to 0.576] | 0.463 [0.006 to 0.921]
  Total number of fibers (Slide II): number analyzed (Participants) | 29 | 15
  Total number of fibers (Slide II) | -24.573 [-59.132 to 9.986] | -22.346 [-64.799 to 20.106]
  Total number of fibers (Slide III): number analyzed (Participants) | 29 | 15
  Total number of fibers (Slide III) | -9.804 [-22.511 to 2.904] | -14.521 [-30.335 to 1.293]
Statistical Analysis 1: Comparison: Givinostat vs Placebo; Fibers with nuclear centralizations (%) at Visit 11; Test type: Superiority; p = 0.1055, ANCOVA — ANCOVA model was performed considering baseline Biopsy histological parameters (Slide I) value as covariate, treatment and concomitant steroid use at baseline as independent class variables; Log Difference of Least Square Means = -0.27, 95% CI 2-sided [-0.59 to 0.06]
Statistical Analysis 2: Comparison: Givinostat vs Placebo; Total number of fibers at Visit 11 (slide II); Test type: Superiority; p = 0.8846, ANCOVA — ANCOVA model was performed considering baseline biopsy histological parameters (Slide II) value as covariate, treatment and concomitant steroid use at baseline as independent class variables; Difference of Least Square Means = -2.23, 95% CI 2-sided [-33.05 to 28.59]
Statistical Analysis 3: Comparison: Givinostat vs Placebo; Total number of fibers (Slide III); Test type: Superiority; p = 0.4054, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Difference of Least Square Means = 4.72, 95% CI 2-sided [-6.62 to 16.06]

8. Secondary Outcome: Mean Change From Baseline to Visit 11 in Percentage for the Biopsy Histology Parameter MFA(%)
Description: Evaluation of histology parameters such as Muscle Fibers Area [MFA](%), were performed comparing muscle biopsies after 12 months of treatment with Givinostat. MFA fraction was determined from biopsies using the mean of available fields. Please note that descriptive statistic data are expressed as least square mean.
Time Frame: after 12 months of treatment (Visit 11)
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of muscle fiber area
Units Other Than Participants: # fields for each biopsy sample
Arm/Group | Givinostat | Placebo
Number analyzed (Participants) | 29 | 15
Number analyzed (# fields for each biopsy sample) | 4 | 4
percentage of muscle fiber area | 0.422 [-10.200 to 11.043] | -2.028 [-16.254 to 12.199]
Statistical Analysis 1: Comparison: Givinostat vs Placebo; Test type: Superiority; p = 0.6340, ANCOVA — [p-value comment as in outcome 7, analysis 1]; Difference of Least Square Means = 2.45, 95% CI 2-sided [-7.87 to 12.77]

9. Secondary Outcome: Mean Change From Baseline to Visit 11 in Percentage for the Biopsy Histology Parameters Adipose Tissue (%)
Description: Evaluation of histology parameters such as Adipose tissue (%) were performed comparing muscle biopsies after 12 months of treatment with Givinostat. Please note that descriptive statistic data are expressed as log least square mean.
Time Frame: after 12 months of treatment (Visit 11)
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of total tissue
Units Other Than Participants: # fields for each biopsy sample
Arm/Group | Givinostat | Placebo
Number analyzed (Participants) | 29 | 15
Number analyzed (# fields for each biopsy sample) | 4 | 4
percentage of total tissue | 0.088 [-0.364 to 0.540] | 0.226 [-0.346 to 0.798]
Statistical Analysis 1: Comparison: Givinostat vs Placebo; Test type: Superiority; p = 0.4893, ANCOVA; Log Difference of Least Square Means = -0.14, 95% CI 2-sided [-0.54 to 0.26]

10. Secondary Outcome: Mean Change From Baseline to Visit 11 in Other Histological Structures
Description: Evaluation of other histological structures like necrotic cells, vessels and any other nonconnective tissue present in the microscopic field were performed comparing muscle biopsies after 12 months of treatment with Givinostat. The value is shown as % compared to the arithmetic mean of the two positive control (i.e., healthy subjects) bands present in the same western blot. Please note that descriptive statistic data are expressed as log least square mean.
Time Frame: after 12 months of treatment (Visit 11)
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of total tissue
Units Other Than Participants: # fields for each biopsy sample
Arm/Group | Givinostat | Placebo
Number analyzed (Participants) | 29 | 15
Number analyzed (# fields for each biopsy sample) | 4 | 4
percentage of total tissue | -0.297 [-0.832 to 0.238] | 0.045 [-0.611 to 0.701]
Statistical Analysis 1: Comparison: Givinostat vs Placebo; Test type: Superiority; p = 0.1498, ANCOVA — This model was performed considering baseline biopsy histological parameters (Slide I) value as covariate, treatment and concomitant steroid use at baseline as independent class variables; Log Difference of Least Square Means = -0.34, 95% CI 2-sided [-0.81 to 0.13]

11. Secondary Outcome: Mean Change From Baseline to Visit 11 in Motor Function Measurement (MFM, Expressed as Log Least Square Mean)
Description: Evaluation were performed using the MFM32 scale, that is a tool designed for neuromuscular diseases and is applicable to all degrees of disease severity. It was validated in terms of reproducibility, construct validity, and concurrent validity. It consists of 32 items (tasks) classified into three dimensions: D1, standing and transfers; D2, axial and proximal motor capacity; and D3, distal motor capacity. Each item is scored on a four-point Likert scale. The generic grading is measured as follows: 0, cannot initiate the task or cannot maintain the starting position; 1, partially performs the task; 2, performs the task with compensatory movements (position maintained for an insufficient period of time, slowness, uncontrolled movements, etc.); and 3, performs the task fully and 'normally', the movement being controlled, mastered, directed, and performed at a constant speed. The overall total score ranging from 0 (severe functional impairment) to 100 (no functional impairment).
Time Frame: after 12 months of treatment (Visit 11)
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Givinostat | Placebo
Number analyzed (Participants) | 34 | 17
score on a scale
  Standing and transfers (D1) | -0.038 [-0.087 to 0.011] | -0.100 [-0.165 to -0.035]
  Axial and proximal motor function (D2) | -0.004 [-0.012 to 0.004] | -0.007 [-0.018 to 0.003]
  Distal motor function (D3) | -0.003 [-0.013 to 0.006] | -0.001 [-0.014 to 0.011]
  Total Score | -0.011 [-0.025 to 0.002] | -0.026 [-0.044 to -0.008]
Statistical Analysis 1: Comparison: Givinostat vs Placebo; Standing and transfers (D1) at Visit 11; Test type: Superiority; p = 0.0602, Mixed Models Analysis — Least squares mean is obtained from the mixed effects model for repeated measures with treatment, visit, visit by treatment interaction and concomitant steroid use at baseline as fixed effect; baseline value is included as a covariate; Log Difference of Least Square Means = 0.06, 95% CI 2-sided [-0.00 to 0.13]
Statistical Analysis 2: Comparison: Givinostat vs Placebo; Axial and proximal motor function (D2) at Visit 11; Test type: Superiority; p = 0.5906, Mixed Models Analysis — [p-value comment as in outcome 11, analysis 1]; Log Difference of Least Square Means = 0.00, 95% CI 2-sided [-0.01 to 0.01]
Statistical Analysis 3: Comparison: Givinostat vs Placebo; Distal motor function (D3) at Visit 11; Test type: Superiority; p = 0.7799, Mixed Models Analysis — [p-value comment as in outcome 11, analysis 1]; Log Difference of Least Square Means = -0.00, 95% CI 2-sided [-0.01 to 0.01]
Statistical Analysis 4: Comparison: Givinostat vs Placebo; Total Score at Visit 11; Test type: Superiority; p = 0.1116, Mixed Models Analysis — [p-value comment as in outcome 11, analysis 1]; Log Difference of Least Square Means = 0.01, 95% CI 2-sided [-0.00 to 0.03]

12. Secondary Outcome: Mean Change From Baseline to Visit 11 in Time Function Test (TFT): Time to Walk/Run 10 Meters
Description: TFT is assessed through 3 different parameters one of which is time to walk/run 10 m. The test was performed with or without orthoses as the patient preferred. He/she was not asked to run, but rather to arrive at the finish line as soon as possible leaving him the choice on how to do so. The assessor walked alongside the patient for safety but couldn't help her/him in any way. The walk/run speed was calculated as 10/time in seconds taken to run/walk 10 m. The test was graded as follows:
  1. Unable to walk independently.
  2. Unable to walk independently but can walk with full leg calipers (KAFOs) or with support of a person.
  3. Highly adapted wide-based lordotic gait. Can't increase walking speed.
  4. Moderately adapted gait. Can pick up speed but can't run.
  5. Able to pick up speed but runs with a double stance phase, i.e., cannot achieve both feet off the ground.
  6. Runs and gets both feet off the ground (with no double stance phase). The higher the grade, the better the outcome.
Time Frame: after 12 months of treatment (Visit 11)
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: sec
Arm/Group | Givinostat | Placebo
Number analyzed (Participants) | 34 | 17
sec | 0.013 [-0.100 to 0.125] | 0.078 [-0.072 to 0.228]
Statistical Analysis 1: Comparison: Givinostat vs Placebo; Time to Walk/Run 10 meters at Visit 11; Test type: Superiority; p = 0.4346, Mixed Models Analysis — [p-value comment as in outcome 11, analysis 1]; Log Difference of Least Square Means = -0.07, 95% CI 2-sided [-0.23 to 0.10]

13. Secondary Outcome: Mean Change From Baseline to Visit 11 in Time Function Test (TFT) Via Time to Climb 4 Standard Steps
Description: TFT is assessed through 3 parameters, one of which is "time to climb 4 standard steps".
  The patient was asked to stand at the bottom of the stairs with his arms by his sides. At the "go" signal, he/she had to walk up the stairs as quickly and safely as possible (using handrails if needed) until reaching an erect position on the top stair. The stair climb speed was calculated as 4/time in seconds taken to climb the 4 standard stairs.
  Grading of the 4-step ascent was:1. Unable to climb 4 stairs.2. Climbs 4 stairs "marking time" (climbs one foot at a time with both feet on a step before moving to next step), using both arms on one or both handrails.3. Climbs 4 stairs "marking time" (idem as up), using one arm on one handrail.4. Climbs 4 stairs "marking time" (idem as up), not needing handrail.5. Climbs 4 stairs alternating feet, needs handrail for support.6. Climbs 4 stairs alternating feet, not needing handrail support.The higher the grade, the better the outcome.
Time Frame: after 12 months of treatment (Visit 11)
Population: Intent-To-Treat Analysis (ITT) Set: all patients assigned treatment by randomization who received at least one dose of study medication. According to the intent to treat principle, patients were analyzed according to the treatment assigned. Efficacy analyses were performed on the ITT set. Please consider the data are showed in Log Least Square Mean
Measure: Least Squares Mean (95% Confidence Interval); unit: sec
Arm/Group | Givinostat | Placebo
Number analyzed (Participants) | 32 | 15
sec | -0.144 [-0.339 to 0.051] | -0.123 [-0.396 to 0.149]
Statistical Analysis 1: Comparison: Givinostat vs Placebo; Time to climb 4 standard steps (sec) at visit 11; Test type: Superiority; p = 0.8914, Mixed Models Analysis; Log Difference of Least Square Means = -0.02, 95% CI 2-sided [-0.32 to 0.28]

14. Secondary Outcome: Mean Change From Baseline to Visit 11 in Time Function Test Via Time to Rise From Floor
Description: Time function test (TFT) is assessed through 3 different parameters, one of which was "time to rise from the floor".
  The patient started the test lying on his back with arms at his sides and was asked to get up as quickly as possible. The rise from floor velocity was calculated as 1/time in seconds taken to stand up. Grading was as follows:
  1. Unable to stand, even with use of a chair.
  2. Assisted Gowers' sign - requires furniture to assist in rising to full upright posture.
  3. Full Gowers' sign - rolls over, stands up with both hands "climbing up" the legs to achieve full upright posture.
  4. Half Gowers' sign - rolls over, stands up with one hand support on leg.
  5. Rolls to the side and/or stands up with one hand or both hands on the floor to start to rise up but does not touch legs.
  6. Stands up without rolling over or using hands. The higher the grade, the better the outcome.
Time Frame: after 12 months of treatment (Visit 11)
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: sec
Arm/Group | Givinostat | Placebo
Number analyzed (Participants) | 29 | 10
sec | 1.392 [-0.968 to 3.753] | 0.774 [-3.014 to 4.562]
Statistical Analysis 1: Comparison: Givinostat vs Placebo; Time to rise from floor at Visit 11; Test type: Superiority; p = 0.7629, Mixed Models Analysis — [p-value comment as in outcome 11, analysis 1]; Difference of Least Square Means = 0.62, 95% CI 2-sided [-3.51 to 4.75]

15. Secondary Outcome: Change From Baseline to Visit 11 in Distance Performed Via 6-minute Walk/Run Test (6MWT, Expressed as Log Least Square Mean)
Description: The 6-minute walk/run test (6MWT) assessed the distance walked in 6 minutes. The 6MWT was performed indoors on a flat, smooth path, at least 30 m long and 3 m wide, with a cone at each end around which the patient had to walk. Six progressively numbered markers were used to mark the distance travelled at each minute. Five progressively lettered markers were used to indicate any falls.
  Two staff members were present during the test; the physiotherapist, to give the patient instructions, and a staff member who followed the patient giving encouragements. The patient was instructed to go from cone to cone as fast as he could but without running, and that he could stop to rest whenever he/she wanted. The time walked, distance walked after each minute, time of each fall and distance walked before each fall were registered.
  A summary of the 6-minute maximum distance walked/run after 12 months of treatment is reported in minutes.
Time Frame: after 12 months of treatment (Visit 11)
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: log [meters]
Arm/Group | Givinostat | Placebo
Number analyzed (Participants) | 34 | 17
log [meters] | -0.058 [-0.118 to 0.002] | -0.046 [-0.128 to 0.036]
Statistical Analysis 1: Comparison: Givinostat vs Placebo; Maximum distance walked after 6 minutes at Visit 11; Test type: Superiority; p = 0.8106, Mixed Models Analysis — [p-value comment as in outcome 11, analysis 1]; Log Difference of Least Square Means = -0.01, 95% CI 2-sided [-0.11 to 0.08]

16. Secondary Outcome: Percentage of Patients With < 10% Worsening in 6MWT After 12 Months of Treatment.
Description: Percentage of patients with < 10% worsening in 6-Minute Walking Test after 12 months of treatment with Givinostat comparing to placebo patients.
Time Frame: after 12 months of treatment (Visit 11)
Population: Intent-To-Treat Analysis (ITT) Set: all patients assigned treatment by randomization who received at least one dose of study medication. According to the intent to treat principle, patients were analyzed according to the treatment assigned. Patients with missing data such that <10% worsening cannot be determined are included in the analysis as having worsened
Measure: Count of Participants; unit: Participants
Arm/Group | Givinostat | Placebo
Number analyzed (Participants) | 34 | 17
Participants | 7 | 1
Statistical Analysis 1: Comparison: Givinostat vs Placebo; <10% worsening at visit 11; Test type: Superiority; p = 0.1626, Cochran-Mantel-Haenszel — P-value is obtained from the two-sided Cochran-Mantel-Haenszel chi-squared test, stratified for concomitant steroid use at baseline

17. Secondary Outcome: Count of Participant Who Lose Ambulation During the Study (From Baseline to Month 12)
Description: Percentage of patients losing the ability to ambulate from baseline to the end of study (Visit 11 or Month 12)
Time Frame: from baseline to the end of month 12
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Givinostat | Placebo
Number analyzed (Participants) | 34 | 17
Participants | 0 | 0

18. Secondary Outcome: Percentage of Patients Who Fell During the 6MWT
Description: A summary of the number of patients who fell and the number of falls occurring during the 6MWT is shown.
Time Frame: after 12 months of treatment (Visit 11)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Givinostat | Placebo
Number analyzed (Participants) | 34 | 17
Participants | 1 | 1

19. Secondary Outcome: Mean Change From Baseline to Visit 11 in Muscle Strength Evaluated by Knee Extension, Elbow Flexion
Description: Evaluation was performed by mean left and right knee extension, mean left and right elbow flexion using the Hand Held Myometry (HHM). Using it, the muscle strength of the knee extensor and elbow flexor were measured via standardized procedures; 3 measurements were recorded from each muscle group on each side. The mean of the 3 measurements was calculated.
  Knee Extension: the pt was sitting, pelvis and knee at a 90° angle. His/her feet were above the ground with the femur in neutral rotation. He/she could hold on to the edge of the bed/chair and, in case, additional stabilization was provided at the distal third of the thigh, just above the knee. The HHM was placed on the anterior surface of the lower third of the tibia, proximal to the ankle joint.
  Elbow flexion: pt lying on his back, arm by his side, elbow flexed at a 90° angle, forearm in supine position. The MMH was placed between the middle and distal third of the forearm, proximal to the radial styloid process.
Time Frame: after 12 months of treatment (Visit 11)
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: Newton
Units Other Than Participants: # of measurements
Arm/Group | Givinostat | Placebo
Number analyzed (Participants) | 34 | 17
Number analyzed (# of measurements) | 3 | 3
Newton
  Left Knee Extension (N): number analyzed (Participants) | 32 | 14
  Left Knee Extension (N) | -1.479 [-10.208 to 7.251] | -5.051 [-15.952 to 5.851]
  Right Knee Extension (N): number analyzed (Participants) | 33 | 16
  Right Knee Extension (N) | 0.703 [-5.212 to 6.618] | -0.460 [-7.705 to 6.784]
  Left Elbow Flexion (N): number analyzed (Participants) | 31 | 14
  Left Elbow Flexion (N) | 1.551 [-10.046 to 13.148] | -2.373 [-17.487 to 12.742]
  Right Elbow Flexion (N): number analyzed (Participants) | 31 | 15
  Right Elbow Flexion (N) | -1.277 [-13.384 to 10.830] | -5.381 [-21.270 to 10.508]
Statistical Analysis 1: Comparison: Givinostat vs Placebo; Left Knee Extension (N) at Visit 11; Test type: Superiority; p = 0.5099, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Difference of Least Square Means = 3.57, 95% CI 2-sided [-7.27 to 14.41]
Statistical Analysis 2: Comparison: Givinostat vs Placebo; Right Knee Extension (N) at Visit 11; Test type: Superiority; p = 0.7355, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Difference of Least Square Means = 1.16, 95% CI 2-sided [-5.73 to 8.06]
Statistical Analysis 3: Comparison: Givinostat vs Placebo; Left Elbow Flexion (N) at Visit 11; Test type: Superiority; p = 0.6037, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Difference of Least Square Means = 3.92, 95% CI 2-sided [-11.22 to 19.06]
Statistical Analysis 4: Comparison: Givinostat vs Placebo; Right Elbow Flexion (N) at Visit 11; Test type: Superiority; p = 0.6178, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Difference of Least Square Means = 4.10, 95% CI 2-sided [-12.35 to 20.55]

20. Secondary Outcome: Mean Changes From Baseline to Visit 11 in Quality of Life (QoL, Assessed by the 36-item Short Form Survey [SF36])
Description: A summary of QoL (SF-36, Single items Short Form survey) in the ITT set is shown.
  QoL (SF-36) is assessed considering:
  * Physical Functioning (PF)
  * Role-Physical (RP)
  * Bodily Pain (BP)
  * General Health (GH)
  * Vitality (VT)
  * Social Functioning (SF)
  * Role-Emotional (RE)
  * Mental Health (MH)
  * Physical Component Summary (PCS)
  * Mental Component Summary (MCS) The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score, the greater the disability. The SF-36 is a set of generic, coherent, and easily administered quality-of-life measures. These measures rely upon patient self-reporting and are widely utilized by managed care organizations for routine monitoring and assessment of care outcomes in adult patients.
Time Frame: after 12 months of treatment (Visit 11)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Givinostat | Placebo
Number analyzed (Participants) | 34 | 17
units on a scale
  Physical Functioning | -1.03 (16.274) | -5.00 (11.989)
  Role-Physical | -2.21 (19.697) | 0.37 (16.006)
  Bodily Pain | 5.12 (19.384) | 2.12 (15.227)
  General Health | 0.82 (14.532) | 1.47 (13.267)
  Vitality | 0.55 (11.654) | 3.68 (12.705)
  Social Functioning | 2.94 (22.415) | 8.82 (20.139)
  Role-Emotional | 0.00 (20.205) | 4.90 (15.607)
  Mental Health | 4.12 (15.997) | 4.41 (13.793)
  Physical Component Summary | -0.17 (5.633) | -1.20 (5.535)
  Mental Component Summary | 1.41 (7.345) | 3.70 (7.177)

21. Secondary Outcome: Number of Patients Experiencing Any Kind of Severity of TEAEs, Serious and Non Serious) From Baseline Through End of Study (EOS).
Description: Treatment-emergent adverse events (TEAEs) are defined as those events with an onset date after study treatment initiation. An AE is an untoward medical occurrence after exposure to a medicine, which is not necessarily caused by that medicine. A serious AE is an adverse reaction that results in death, is life-threatening, requires hospitalisation or prolongation of existing hospitalisation, results in persistent or significant disability or incapacity, or is a birth defect.
Time Frame: Throughout the study, till week 52 +/-7 days
Population: Safety Set: all patients who received at least one dose of study medication. Patients were analyzed according to the study treatment actually received. The safety set was used for the safety analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Givinostat | Placebo
Number analyzed (Participants) | 34 | 17
Participants
  Number of patients with any TEAEs | 30 | 9
  Number of patients with serious TEAEs | 0 | 0
  Number of patients with TEAEs leading to interruption of study treatment | 11 | 1
  Number of patients with fatal TEAEs | 0 | 0
  Number of patients with mild TEAEs | 30 | 9
  Number of patients with moderate TEAEs | 12 | 1
  Number of patients with severe TEAEs | 5 | 0
  Number of patients with TEAEs related to study treatment | 29 | 4
  Number of patients with TEAEs not related to study treatment | 25 | 8

22. Secondary Outcome: Mean Change From Baseline to Visit 11 in the Percentage of Fat Fraction of Lower Limb Muscles (Log)
Description: as for outcome 3
Time Frame: after 12 months of treatment (at Visit 11)
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: log[percentage of fat in muscle]
Units Other Than Participants: MRI images for each timepoint
Arm/Group | Givinostat | Placebo
Number analyzed (Participants) | 34 | 17
Number analyzed (MRI images for each timepoint) | 5 | 5
log[percentage of fat in muscle] | 0.012 [-0.017 to 0.041] | 0.038 [0.003 to 0.073]
Statistical Analysis 1: Comparison: Givinostat vs Placebo; Medial Thigh at visit 11; Test type: Superiority; p = 0.1165, ANCOVA — ANCOVA model was performed considering baseline fat fraction of lower limb muscles value as covariate and treatment and concomitant steroids use at baseline as independent class variables; log difference of Least Square Means = -0.03, 95% CI 2-sided [-0.06 to 0.01]

23. Secondary Outcome: Mean Change From Baseline to Visit 11 in Contractile Area of Lower Limb Muscles (MRI) (Log)
Description: as for outcome 5
Time Frame: after 12 months of treatment
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: centimeters^2
Units Other Than Participants: MRI muscle images for each timepoint
Arm/Group | Givinostat | Placebo
Number analyzed (Participants) | 34 | 17
Number analyzed (MRI muscle images for each timepoint) | 5 | 5
centimeters^2 | 0.025 [-0.042 to 0.092] | -0.022 [-0.104 to 0.059]
Statistical Analysis 1: Comparison: Givinostat vs Placebo; Hamstrings at Visit 11; Test type: Superiority; p = 0.1939, ANCOVA — ANCOVA model was performed considering baseline CSA as covariate and treatment and concomitant steroids use at baseline as independent class variables; Log difference of Least Square Means = 0.05, 95% CI 2-sided [-0.02 to 0.12]

24. Secondary Outcome: Mean Change From Baseline to Visit 11 in Biopsy Histology Parameters: CSA by Type (I or II Fibers), Total CSA (Log)
Description: as for outcome 6
Time Frame: After 12 months of treatment (Visit 11)
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: log [micrometers^2]
Units Other Than Participants: # fields for each biopsy sample
Arm/Group | Givinostat | Placebo
Number analyzed (Participants) | 34 | 17
Number analyzed (# fields for each biopsy sample) | 4 | 4
log [micrometers^2] | 0.255 [-0.069 to 0.579] | 0.246 [-0.166 to 0.658]
Statistical Analysis 1: Comparison: Givinostat vs Placebo; CSA Type I; Test type: Superiority; p = 0.9493, ANCOVA — ANCOVA model was performed considering baseline biopsy histological parameters (slide III) value as covariate, treatment and concomitant steroids use at baseline as independent class variables; Log difference of Least Square Means = 0.01, 95% CI 2-sided [-0.29 to 0.30]

25. Secondary Outcome: Mean Change From Baseline to Visit 11 in Percentage for the Following Histology Parameters: Fibers With Nuclear Centralizations (%), Total Number of Fibers (%), Regenerative Fibers (%). (Log)
Description: as for outcome 7
Time Frame: after 12 months of treatment (Visit 11)
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: log[percentage of fibers]
Units Other Than Participants: # fields for each biopsy sample
Arm/Group | Givinostat | Placebo
Number analyzed (Participants) | 34 | 17
Number analyzed (# fields for each biopsy sample) | 4 | 4
log[percentage of fibers]
  Total number of fibers (Slide I) | -0.207 [-0.446 to 0.032] | -0.257 [-0.552 to 0.037]
  Regenerative fibers | 0.667 [-0.031 to 1.365] | 1.104 [0.248 to 1.961]
Statistical Analysis 1: Comparison: Givinostat vs Placebo; Total number of Fibers at Visit 11 (slide I); Test type: Superiority; p = 0.6265, ANCOVA — ANCOVA model was performed considering baseline biopsy histological parameters (slide I) value as covariate, treatment and concomitant steroids use at baseline as independent class variables; Log difference of Least Square Means = 0.05, 95% CI 2-sided [-0.16 to 0.26]
Statistical Analysis 2: Comparison: Givinostat vs Placebo; Regenerative Fibers (%) at Visit 11; Test type: Superiority; p = 0.1562, ANCOVA — ANCOVA model was performed considering baseline biopsy histological parameters (slide II) value as covariate, treatment and concomitant steroids use at baseline as independent class variables; Log difference of Least Square Means = -0.44, 95% CI 2-sided [-1.05 to 0.17]

ADVERSE EVENTS:
Time Frame: Throughout the study, from screening (visits 1 and 2) to EOS/early withdrawal (V11, at week 48 ± 7 days) till follow-up visit (visit 12, at week 52 ± 7 days). This means the AEs were monitored from screening to day 364 ± 7.
Description: Patients who completed the study (12 months of treatment) were asked to return to the center for the Follow-up visit 4 weeks after the last dose of study treatment (4 weeks ±1). However, a patient that was discontinued from the study treatment was asked to return for the early withdrawal visit within 4 weeks of the last dose of study treatment.
Groups:
- Givinostat: Givinostat oral suspension (10 mg/mL) twice daily in a fed state
  givinostat: suspension of givinostat (10 mg/mL) bid
Arm/Group | Givinostat | Placebo
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/17
Other Adverse Events (participants affected / at risk) | 30/34 | 9/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Givinostat (N=34) | Placebo (N=17)
Lymphocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 16 (16) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 1 (1)
Hyperpyrexia (General disorders) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 2 (2) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Chest injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tooth injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 1 (1)
Blood phosphorus increased (Investigations) | 0 (0) | 1 (1)
Blood potassium increased (Investigations) | 0 (0) | 1 (1)
Blood sodium increased (Investigations) | 0 (0) | 1 (1)
Blood triglycerides increased (Investigations) | 4 (4) | 1 (1)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 1 (1)
Heart rate increased (Investigations) | 2 (2) | 0 (0)
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 17 (20) | 0 (0)
Weight increased (Investigations) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 10 (10) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle hypertrophy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0)
Hand-arm vibration syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Tooth repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Umbilical hernia repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Epistaxis (Vascular disorders) | 1 (1) | 0 (0)
Haematuria (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-06-20): https://cdn.clinicaltrials.gov/large-docs/35/NCT03238235/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-27): https://cdn.clinicaltrials.gov/large-docs/35/NCT03238235/SAP_001.pdf